CLINICAL TRIAL: NCT05221853
Title: Comparison of Standard Breath-hold Cardiac MRI With a Faster, Free-breathing Scan
Brief Title: Real-time MRI for Evaluating Cardiac Volumetry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 0768; 270285 (Other: Health Research Authority)
Record Dates: First submitted 2021-11-15; First posted 2022-02-03 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Left Ventricle Abnormality

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: cardiovascular magnetic resonance — CMR scan at 3 Tesla

SUMMARY:
This study will compare the accuracy of a real-time Cine sequence in assessing cardiac volumetry.

DETAILED DESCRIPTION:
This is a single-centre prospective study involving up to 570 patients with known or suspected cardiac disease referred for routine clinical cardiovascular magnetic resonance (CMR) assessment at Glenfield General Hospital, Leicester. In addition to standard multi-breath-hold steady-state free precession (SSFP) imaging (undertaken as part of the routine scan), each patient will also undergo additional imaging with a non-breath-hold multi-slice real-time cine sequence.

The primary outcome is the assessment of cardiac volumetry and function (end-diastolic volume, end-systolic volume, stroke volume, ejection fraction and myocardial mass) as measured by (1) the standard multi-breath-hold SSFP technique and (2) the non-breath-hold multi-slice real-time cine sequence. Secondary outcome measures will be (1) the time required for each scan, and (2) image quality for each scan. An additional secondary outcome will be to compare indexed cardiac volumes with those indexed according to measured body-surface area.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥ 18 years
2. Referred for routine CMR imaging
3. Willing and able to give informed consent
4. Willing and able to comply with the requirements of the study
5. Able to understand written English

Exclusion Criteria:

1. Severe claustrophobia
2. Absolute contraindications to CMR (those with CMR conditional or safe devices will be eligible for inclusion)
3. Unable to provide informed consent
4. Participants unable to understand written English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults patients referred for routine cardiac MRI at Glenfield Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 570 (Estimated)
Dates: Start 2021-02-23 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Cardiac volumetric assessment 1 | 1 day
  Left ventricular ejection fraction
Cardiac volumetric assessment 2 | 1 day
  Left ventricular end-diastolic volume
Cardiac volumetric assessment 3 | 1 day
  Left ventricular myocardial mass
Cardiac volumetric assessment 4 | 1 day
  Right ventricular ejection fraction
Cardiac volumetric assessment 5 | 1 day
  Right ventricular end-diastolic volume
Cardiac strain assessment 1 | 1 day
  Left ventricular global longitudinal strain
Cardiac strain assessment 2 | 1 day
  Left ventricular global circumferential strain

SECONDARY OUTCOMES:
Time | 1 day
  the time required for each scan under evaluation (real-time Cine and standard Cine)
Image quality assessment | 1 day
  Image quality of each scan component, assessed visually on a 4-point score - excellent (3), good (2), moderate (1) and poor (0).
Body-surface area | 1 day
  planimetered body-surface area

CONTACTS AND LOCATIONS:
Overall Officials: Jayanth Arnold, Principal Investigator — University of Leicester
Locations (1):
- Glenfield Hospital, Leicester, Leics, United Kingdom

IPD SHARING:
Plan to Share IPD: No
no plan to share data

REFERENCES:
- [Derived] Elshibly M, Shergill S, Parke K, Budgeon C, England R, Grafton-Clarke C, Elshibly F, Kellman P, McCann GP, Arnold JR. Standard breath-hold versus free-breathing real-time cine cardiac MRI-a prospective randomized comparison in patients with known or suspected cardiac disease. Eur Heart J Imaging Methods Pract. 2025 Apr 25;3(1):qyaf042. doi: 10.1093/ehjimp/qyaf042. eCollection 2025 Jan. PMID 40308862